CLINICAL TRIAL: NCT07259512
Title: Comparative Effects of Single Versus Twice-Daily Ramipril Dosing on Renal Function in Patients With Chronic Kidney Disease and Heart Failure With Reduced Ejection Fraction: Evaluation of Plasma Renin Activity, Malondialdehyde, Interleukin-6, Albuminuria, and Cystatin C
Brief Title: Single and Twice-daily Dosing of Ramipril on Renal Function in Chronic Kidney Disease Patients With Reduced Ejection Fraction Heart Failure
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Evi Liliek Wulandari (Other)
Responsible Party: Sponsor-Investigator, Evi Liliek Wulandari, Principal Investigator, Consultant Internist (Internal Medicine Specialist), Universitas Sebelas Maret
Organization: Universitas Sebelas Maret (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 041/UN27.46/TA.04.19/KEP/EC/20
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease; Heart Failure With Reduced Ejection Fraction (HFrEF)
Keywords: Chronic Kidney Disease; HFrEF; Ramipril
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Ramipril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in parallel to one of two treatment groups: once-daily ramipril (10 mg every 24 hours) or twice-daily ramipril (5 mg every 12 hours). Each participant remains in the same assigned arm for the entire 30-day treatment period, and outcomes are assessed at baseline and day 30.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Once-Daily Ramipril (Experimental): Participants receive ramipril 10 mg once daily for 30 days
  Interventions: Drug: Ramipril
- Twice-Daily Ramipril (Experimental): Participants receive ramipril 5 mg twice daily for 30 days
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril — Ramipril administered either as 10 mg once daily or 5 mg twice daily for 30 days
  Other Names: ACE inhibitor

SUMMARY:
This study compares the effects of once-daily versus twice-daily ramipril dosing on renal function in chronic kidney disease (CKD) patients with heart failure with reduced ejection fraction (HFrEF). Outcomes include changes in plasma renin activity, malondialdehyde, interleukin-6, albuminuria, and cystatin C after 30 days of therapy.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) frequently coexists with heart failure with reduced ejection fraction (HFrEF), characterized by neurohormonal activation, inflammation, oxidative stress, and progressive renal deterioration. Activation of the renin-angiotensin-aldosterone system (RAAS) contributes significantly to both renal and cardiac dysfunction. Ramipril, an ACE inhibitor, is widely recommended for CKD with albuminuria and HFrEF. However, discrepancies exist in guidelines regarding once-daily versus twice-daily administration. These differences may influence RAAS suppression effectiveness and patient adherence.

This randomized, double-blind, parallel assignment clinical trial investigates the impact of once-daily (10 mg every 24 hours) versus twice-daily (5 mg every 12 hours) ramipril dosing on renal biomarkers in CKD patients with HFrEF. Outcomes include plasma renin activity (PRA), malondialdehyde (MDA), interleukin-6 (IL-6), albuminuria, and cystatin C measured over a 30-day treatment period. The study aims to provide scientific evidence to support optimal ramipril dosing strategies that improve renal outcomes among patients with CKD and reduced ejection fraction heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male with age >18 years old
* Patients with a diagnosis of CKD stage 3-5 non-dialysis with low ejection fraction heart failure (ejection fraction < 40%)

Exclusion Criteria:

* Receiving hemodialysis therapy
* History of intolerance to ACE inhibitors
* Refractory hyperkalemia
* Pregnancy
* History of angioedema to ACE inhibitors
* Receiving sacubitril-valsartan therapy
* Receiving ARB therapy
* Hypotension with blood pressure <90/60, or patients in shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Plasma Renin Activity (PRA) | 30 days
  Change in plasma renin activity from baseline to day 30.
Change in Malondialdehyde (MDA) | 30 days
  Change in plasma MDA levels as a biomarker of oxidative stress
Change in Interleukin-6 (IL-6) | 30 days
  Change in serum IL-6 levels as a marker of systemic inflammation
Change in Albuminuria | 30 days
  Change in albumin-creatinine ratio (ACR) from baseline to day 30
Change in Cystatin C | 30 days
  Change in serum cystatin C levels as a marker of glomerular filtration

SECONDARY OUTCOMES:
Change in Serum Creatinine | 30 days
  Change in serum creatinine concentration from baseline to day 30, measured by standard hospital laboratory methods
Change in Estimated Glomerular Filtration Rate (eGFR) | 30 days
  Change in estimated glomerular filtration rate (eGFR) from baseline to day 30, calculated using the CKD-EPI equation
Change in Blood Pressure (Systolic and Diastolic) | 30 days
  Change in clinic-measured systolic and diastolic blood pressure from baseline to day 30
Incidence of Treatment-Related Adverse Events | 30 days
  Number and type of adverse events considered related to ramipril during 30 day treatment period (e.g. hyperkalemia), graded by severity

CONTACTS AND LOCATIONS:
Locations (1):
- UNS Hospital, Kartasura, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kidney Disease: Improving Global Outcomes (KDIGO) Diabetes Work Group. KDIGO 2020 Clinical Practice Guideline for Diabetes Management in Chronic Kidney Disease. Kidney Int. 2020 Oct;98(4S):S1-S115. doi: 10.1016/j.kint.2020.06.019. No abstract available. PMID 32998798
- [Result] Ariton DM, Jimenez-Balado J, Maisterra O, Pujadas F, Soler MJ, Delgado P. Diabetes, Albuminuria and the Kidney-Brain Axis. J Clin Med. 2021 May 27;10(11):2364. doi: 10.3390/jcm10112364. PMID 34072230
- [Result] Kreiner FF, Kraaijenhof JM, von Herrath M, Hovingh GKK, von Scholten BJ. Interleukin 6 in diabetes, chronic kidney disease, and cardiovascular disease: mechanisms and therapeutic perspectives. Expert Rev Clin Immunol. 2022 Apr;18(4):377-389. doi: 10.1080/1744666X.2022.2045952. Epub 2022 Mar 1. PMID 35212585
- [Result] Jakopin E, Knehtl M, Hojs NV, Bevc S, Piko N, Hojs R, Ekart R. Treatment of acute kidney injury with continuous renal replacement therapy and cytokine adsorber (CytoSorb(R)) in critically ill patients with COVID-19. Ther Apher Dial. 2024 Dec;28(6):941-950. doi: 10.1111/1744-9987.14182. Epub 2024 Jul 3. PMID 38958006
- [Result] Nijst P, Verbrugge FH, Martens P, Bertrand PB, Dupont M, Francis GS, Tang WW, Mullens W. Plasma renin activity in patients with heart failure and reduced ejection fraction on optimal medical therapy. J Renin Angiotensin Aldosterone Syst. 2017 Jul-Sep;18(3):1470320317729919. doi: 10.1177/1470320317729919. PMID 28875746
- [Result] Arifiyanto, A. Y., Dwi Laksono, A., Chalidyanto, D., Taniasari, N., & Kusumaningtyas, W. (2021). Factors Related to the Prevalenceof Chronic Kidney Disease in Indonesia:An Ecological Study. Indian Journal of Forensic Medicine & Toxicology, 15(3), 1867-1873.
- [Result] Tedeschi A, Agostoni P, Pezzuto B, Corra' U, Scrutinio D, La Gioia R, Raimondo R, Passantino A, Piepoli MF. Role of comorbidities in heart failure prognosis Part 2: Chronic kidney disease, elevated serum uric acid. Eur J Prev Cardiol. 2020 Dec;27(2_suppl):35-45. doi: 10.1177/2047487320957793. PMID 33238740

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT07259512/Prot_SAP_ICF_001.pdf